CLINICAL TRIAL: NCT00069693
Title: Clinical Laboratory Evaluation of Chronic Orthostatic Intolerance
Brief Title: Evaluation of Chronic Orthostatic Intolerance
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030314; 03-N-0314
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-05

CONDITIONS: Syncope
Keywords: Dysautonomia; Sympathetic Nervous System; Autonomic Nervous System; Syncope; Post Tachycardia Syndrome; POTS; Neurocardiogenic Syncope; Baroreflex; Norepinephrine; Epinephrine; Neurocardiology; Chronic Orthostatic Intolerance; COI; Healthy Volunteer; HV
MeSH Terms: conditions — Syncope; Autonomic Nervous System Diseases; Syncope, Vasovagal

SUMMARY:
This study will conduct tests with patients with primary chronic orthostatic intolerance (COI) to learn more about this disorder of the autonomic nervous system.

Healthy normal volunteers and patients 18 years of age and older with COI may be eligible for this study. Participants undergo one or more of the following tests and procedures:

* Blood studies, including arterial catheter insertion to measure blood pressure and collect arterial blood samples, blood flow studies using sensors applied to the skin and a pressure cuff around a limb, blood volume studies using injection of radioactively labeled human serum albumin and gene studies to look for genetic abnormalities associated with certain proteins.
* Imaging studies, including CT scan of the adrenal glands, heart ultrasound, and PET scanning.
* Electrocardiogram
* Microdialysis to measures levels of chemicals in the body fluid of certain tissues. A thin tube is inserted into the skin and a solution is passed through it. Chemicals in the body tissues enter the solution in the tube. The solution is collected and the chemical levels are measured.
* Neck suction. Neck suction is applied to test a reflex the brain uses to regulate blood pressure.
* Perometry. Limb volume is measured using an infrared light that moves up the limb.
* Quantitative sudomotor axon reflex test to evaluate an aspect of autonomic nervous system function. A small amount of a brain chemical (acetylcholine) is applied to the skin with a tiny amount of electricity, and the sweat in a nearby patch of skin is measured.
* Skin electrical conduction test using sensors on the skin to measure sweat production.
* Skin and core temperature measurements using sensors on the skin and in the ear canal.
* Tilt table test. The subject lies on a table, secured with straps around the chest and legs. Sensors are placed on the arms and chest to monitor blood pressure, pulse rate, and heart rhythm. A catheter is placed in a vein in each arm to collect blood samples and give drugs. Another catheter is placed in an artery to draw blood and monitor blood pressure. The subject is given an infusion of norepinephrine and epinephrine, and baseline measures and blood samples are taken. The table is tilted upright and more measurements and blood samples are taken at intervals for up to 30 minutes. The table is returned to a horizontal position and additional measurements and samples may be taken.

Drugs may be administered during the tests, including acetylcholine, epinephrine, and norepinephrine, radioactive chemicals used in imaging studies, and drugs that affect blood vessels, heart rate, and force of heart contractions.

DETAILED DESCRIPTION:
This protocol is to identify and characterize distinct types of chronic orthostatic intolerance (COI). COI can be a manifestation of primary chronic autonomic failure, which is covered under a separate protocol. The present protocol concerns patients with COI who under resting conditions have intact sympathetic neurocirculatory function. COI can reflect different pathophysiologic mechanisms; until now, few studies have attempted to distinguish these mechanisms in individual patients. We hypothesize that results of clinical assessment and physiologic, chemical, pharmacologic, and imaging tests will reveal internally consistent patterns that distinguish particular forms of COI. We wish to determine the relative frequencies of these forms in a referral population. The first phase of testing is to identify sympathetic neurocirculatory failure, baroreflex failure, and secondary causes of COI (hypovolemia, excessive orthostatic venous pooling, or excessive orthostatic extravasation). In a subsequent inpatient phase, tilt table testing is done, with concurrent hemodynamic and chemical measurements, to confirm subtypes of postural tachycardia syndrome and neurocardiogenic syncope. The results of these evaluations will be used for stratification of specific, pathophysiologically defined diagnostic groups for therapeutic protocols. In an off-site study, we will evaluate members of a large family where COI seems to be transmitted as an autosomal dominant trait.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects are patients with COI and adult healthy volunteers of similar age, gender, and body mass.

Participation in this protocol is offered to people 18 years old or older, independently of gender, race, age, ethnicity, religion, or any other demographic or sociopolitical classifications.

The subjects in the second off-site study are family members of the identified proband. Participation in this protocol is offered to people 18 years old or older, independently of gender, race, ethnicity, religion, or any other demographic or sociopolitical classifications.

In the second off-site study, participation is also offered to subjects 10 to 17 years old, provided that appropriate informed consent/assent has been given by the subject and his/her parent or guardian.

EXCLUSION CRITERIA:

Age: Minors younger than 18 years old are excluded, except for the off-site study. Advanced age does not constitute an exclusion criterion. For subjects more than 55 years old, carotid Doppler studies are done, and subjects with significant carotid disease (stenosis by atherosclerosis) are excluded. In the off-site study, minors younger than 10 years old are excluded. For the second off-site study, minors younger than 10 years old are excluded. Advanced age does not constitute an exclusion criterion. Except for the second off-site study, people less than 18 years old are excluded.

Risk: A candidate subject is excluded if, in the judgment of the Principal Investigator or Clinical Director, protocol participation would place the subject at substantially increased acute medical risk. This includes the risks associated with air travel to the NIH. A candidate subject is excluded if, in the opinion of the Principal Investigator or Clinical Director, the medical risk outweighs the potential scientific benefit.

Disqualifying Conditions: A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are hepatic or renal failure, a history of tachyarrhythmias, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, symptomatic coronary heart disease, diabetes mellitus, hyperthyroidism, and allergy or sensitivity to iodinated contrast media or any of the planned drugs. A positive HIV rest result does not necessarily exclude a patient from participating.

Medications: A candidate subject is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Examples are tricyclic antidepressants, anticoagulants, beta-adrenoceptor blockers, phenothiazines, barbiturates, monoamine oxidase inhibitors, acetaminophen, and alpha-adrenoceptor agonists or antagonists. Patients on one or more of these drugs are not excluded, if the drugs are tapered and discontinued before undergoing the clinical laboratory testing. Patients are not to discontinue any medications before the patient or the patient's doctor discusses this with the Principal Investigator. If it is decided that discontinuing medications would be unsafe, then the patient is excluded from the study. Patients with known or suspected allergy or hypersensitivity to any test drug are excluded. Patients unable to discontinue nicotine or alcohol for 24 hours prior to evaluation are excluded.

Patients with chronic orthostatic intolerance often take several medications that could interfere with the scientific results of this protocol. Temporary discontinuation of medications as outpatients, even with the approval of the referring physician, introduces some risk. To maximize patient safety, we may admit patients for monitoring as inpatients while medications are tapered or stopped.

In the second off-site study, subjects are tested while on their usual medications.

Herbal Medicines and Dietary Supplements: Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate. Subjects in the off-site study may continue their herbal medicines or dietary supplements.

Practical Limitations: Patients in whom we feel it would be difficult to insert a catheter into a vein are excluded. Subjects who are not expected clinically to tolerate lying still during the procedures are excluded. In the second off-site study, if an i.v. cannot be placed, or the subject refuses to have an i.v. placed then a DNA sample may be obtained by buccal smear or obtaining saliva.

Pregnancy: Pregnant or lactating women are excluded. In the second off-site study, pregnancy is not an exclusion criterion.

The Investigators may also exclude a subject from further participation, such as in the event of known or suspect falsification of medical history information or refusal to undergo planned tests or procedures, without loss of benefits to which the subject was previously entitled.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2003-09-26; Study Completion 2008-08-05

CONTACTS AND LOCATIONS:
Locations (3):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Canada (2):
  - Hospital Sacre-Coeur de Montreal, Montreal
  - University of Ottawa Heart Institute, Ottawa

REFERENCES:
- [Background] Robertson D. The epidemic of orthostatic tachycardia and orthostatic intolerance. Am J Med Sci. 1999 Feb;317(2):75-7. doi: 10.1097/00000441-199902000-00001. No abstract available. PMID 10037110
- [Background] Goldstein DS, Holmes C, Frank SM, Dendi R, Cannon RO 3rd, Sharabi Y, Esler MD, Eisenhofer G. Cardiac sympathetic dysautonomia in chronic orthostatic intolerance syndromes. Circulation. 2002 Oct 29;106(18):2358-65. doi: 10.1161/01.cir.0000036015.54619.b6. PMID 12403667
- [Background] Furlan R, Jacob G, Snell M, Robertson D, Porta A, Harris P, Mosqueda-Garcia R. Chronic orthostatic intolerance: a disorder with discordant cardiac and vascular sympathetic control. Circulation. 1998 Nov 17;98(20):2154-9. doi: 10.1161/01.cir.98.20.2154. PMID 9815870